CLINICAL TRIAL: NCT06802094
Title: Case-Control Research of the Movement Strategies Used During Balance Tasks in Children With and Without Developmental Coordination Disorder
Brief Title: Movement Strategies During Balance Tasks in Children With and Without Developmental Coordination Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Katrijn Klingels, Principal investigator, Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: B1152024000023
Record Dates: First submitted 2025-01-27; First posted 2025-01-30 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Development Coordination Disorder; Typical Developed Children
Keywords: Postural control; Movement strategies; Brain activity; Postural balance [Mesh]; Pediatrics [Mesh]; Motor Skills Disorders [Mesh]
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Intervention Model Description: Case-control study (Children with and without Developmental Coordination Disorder) with a follow-up measurement for retention and transfer after one week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Learning of a new balance task in virtual reality (Experimental): All children will perform a single training session (30 minutes) in a virtual reality environment, where one game will be played to challenge their balance. After one week, the children will play two games in the virtual reality environment to look at the retention (same game as first session) and transfer (similar game as first session).
  Interventions: Other: Single-session balance intervention in virtual reality

INTERVENTIONS:
Other: Single-session balance intervention in virtual reality — Single-session balance intervention (30 minutes) in a virtual reality environment, the Gait Real-time analysis Interactive Lab (GRAIL) or the Computer Assisted Rehabilitation Environment (CAREN) in children with and without Developmental Coordination Disorder (Motek Medical, The Netherlands).

SUMMARY:
The main objective of the study is to gain insights in how children learn a balance task and whether there is a difference between children with and without Developmental Coordination Disorder. Furthermore, the investigators are interested in the brain activity of these children while learning this new balance task.

ELIGIBILITY:
Inclusion Criteria:

For children with DCD

* Children with the clinical diagnosis of Developmental Coordination Disorder (DCD) based on criteria of the DSM-5 (APA, 2013), diagnosed by a pediatrician.
* Children who have no formal diagnosis are evaluated by the research team using the diagnostic criteria as outlined in the inclusion criteria, these children will be included as "suspected of having DCD"
* Balance problems need to be present and objectified with the Balance Evaluation Systems Test for Children, second edition (Kids-BESTest-2). (total score below 80%)

For children without DCD

* Total score at or below the 25th percentile on the Movement Assessment Battery for children, second edition
* Normal postural control, objectified by the Kids-BESTest-2 (score at or above 80%)
* Match with children with DCD based on their sex, age and potential comorbidities.

Exclusion Criteria:

Presence of:

* Intellectual problems
* Visual problems
* Vestibular problems
* Neurological conditions
* Not able to follow instructions due to behavioral problems
* Refuse to participate

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Changes in the center of mass velocity and acceleration after a single-training session in VR and after a one-week retention | Baseline, after 30 minutes intervention, one week
  Measurement of the movement strategies used by children with and without Developmental Coordination Disorder (DCD) during a balance task. The movement strategies are measured by looking at the center of mass velocity and acceleration during this balance task. The goal is to: (1) investigate whether there is a difference in the used strategies between baseline and after a single training session of 30 minutes; (2) see whether the changes stay present after a one-week retention; (3) see whether there are differences between children with and without DCD.

SECONDARY OUTCOMES:
Hemodynamic response in cortical brain regions during balance tasks | Baseline, one week
  Measurement of the changes in Oxy- and Deoxyhemoglobin concentrations (μmol/l) (baseline vs task condition), with the use of Functional Near-Infrared Spectroscopy (fNIRS), during the execution of balance tasks. The regions of interest are determinded based on the evidence of brain areas needed for postural control tasks in healthy individuals, and affected brain regions in children with DCD in a variety of tasks (frontal and parietal regions).
  The goal is to: (1) determine whether brain activity patterns can be an explanation of the movement strategies used during the single-training session; (2) determine the test-retest reliability of fNIRS during balance tasks in children.
  The NIRSport 2 (NIRx Medical Technologies, GE) with continuous wave imaging (760nm;850nm) is used.
Score on a comprehensive postural control measurement, Kids-BESTest-2 | Baseline
  Score on the Balance Evaluation Systems Test for Children, second edition. The test consists of 6 domains. A score below 80% is the cut-off which corresponds to a postural control problem. The scores give an idea in which domain of postural control the problems are present.

OTHER OUTCOMES:
Score on a general motor scale, Movement Assessment Battery for Children, second edition | Baseline
  The MABC-2 consists of 3 domains (manual dexterity, aiming and catching, balance) with a total of 8 tasks. The test gives a general idea about the motor develompment of children on different domains.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasselt Univeristy, Faculty of Rehabilitation Sciences, Diepenbeek, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided